CLINICAL TRIAL: NCT01103674
Title: Feasibility Study For Safety and Efficacy Evaluation Of The Combined Ablation Procedure For The Treatment Of Drug Refractory Symptomatic Paroxysmal Atrial Fibrillation
Brief Title: Safety and Efficacy Study of the Combined Ablation Procedure to Treat Paroxysmal Atrial Fibrillation
Acronym: CAP STOPS AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment challenges, only one patient enrolled
Sponsor: nContact Surgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAL-1150
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2012-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; AF; Atrial Fibrillation; RF ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Numeris-AF Guided Coagulation System (Other)
  Interventions: Device: Numeris®-AF Guided Coagulation System with VisiTrax®

INTERVENTIONS:
Device: Numeris®-AF Guided Coagulation System with VisiTrax® — Combined epicardial / endocardial procedure using the Numeris®-AF Guided Coagulation System with VisiTrax® epicardially and the Biosense Webster ThermoCool Catheter in conjunction with the Carto Navigation System endocardially.

SUMMARY:
This is a multi-center, prospective, open label, feasibility clinical study,evaluating the safety and efficacy of the combined ablation procedure for the treatment of symptomatic paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to evaluate the safety and efficacy of the epicardial / endocardial combined procedure for the treatment of drug refractory symptomatic Paroxysmal Atrial Fibrillation (AF) patients, using the nContact Numeris®-AF Guided Coagulation System with VisiTrax® epicardially and the Biosense Webster NaviStar® ThermoCool® Diagnostic/Ablation deflectable Tip Catheter in conjunction with the Carto Navigation System endocardially.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years; < 80 years
* Left atrium less than or equal to 6.5 cm (TTE)
* Symptomatic paroxysmal AF
* Provided written informed consent
* Refractory to at least one AAD (class I, II, III or IV)

Exclusion Criteria:

* Patients requiring concomitant surgery
* Left ventricular ejection fraction < 30%
* Pregnant or planning to become pregnant during study
* Co-morbid medical conditions that limit one year life expectancy
* Measured left ventricular wall thickness > 1.5 cm
* History of coagulopathy
* Previous cardiac surgery
* Right ventricular outflow tract obstruction
* History of pericarditis
* Previous cerebrovascular accident (CVA), excluding fully resolved TIA
* Patients who have severe chronic obstructive pulmonary disease (COPD)
* Patients who have an active infection or sepsis
* Patients who have uncorrected reversible cause(s) of AF
* Patients who are contraindicated for anticoagulants
* Patients who are being treated for arrhythmias other than AF
* Patients who have had any previous AF or left atrial catheter ablation
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment.
* Not competent to legally represent him or herself (e.g., requires a guardian or caretaker as a legal representative).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
AF free off all Class I and III Anti Arrhythmic Drugs (AADs). | 12 months
  The primary efficacy data will be an evaluation of the number of subjects free from AF and free of all Class I and III Anti Arrhythmic Drugs (AADs) from 3 months through 12 months post procedure.

SECONDARY OUTCOMES:
AF free regardless of the Class I and III AADs status | 12 months
  The secondary efficacy data will be an evaluation of the number of subjects free from AF regardless of their Class I and III AADs status from 3 months through 12 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Horton, MD, Principal Investigator — Texas Cardiac Arrhythmia Institute, St. David's Medical Center
Locations (2):
- United States (2):
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Texas Cardiac Arrhythmia Institute, St. David's Hospital, Austin, Texas